CLINICAL TRIAL: NCT00787501
Title: Imaging Antidepressant vs. Cognitive Behavior Therapy Effects on Unipolar Depression
Acronym: ssrifMRI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: The Pittsburgh Foundation (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Greg Siegle, Associate Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO07100326; M2007-0114; R01MH074807 (NIH)
Record Dates: First submitted 2008-11-05; First posted 2008-11-07 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression; Selective Serotonin Reuptake Inhibitors; Cognitive Behavior Therapy; Cognitive Therapy; antidepressant medications
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Escitalopram; Fluoxetine; Sertraline; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SSRIs (Active Comparator): Selective Serotonin Reuptake Inhibitors
  Interventions: Drug: SSRI
- CBT (Active Comparator): Cognitive Behavior Therapy
  Interventions: Behavioral: CBT

INTERVENTIONS:
Drug: SSRI — SSRI: 25 patients will receive 14 weeks of an FDA approved selective serotonin reuptake inhibitor (SSRI), administered under the supervision of a staff psychiatrist. After an initial 30-45 minute session patients will be seen for 15-30 minute sessions for 16-20 sessions over 14 weeks. Medication will begin with 10mg escitalopram daily (or its equivalent), increased to 30 mg/day (or its equivalent) by week 6 if pt has not achieved a minimum level of response (i.e., CGI < 2) and tolerability is adequate. Nonresponse at week 10 (CGI < 2) will be cause for medication switch or augmentation.
  Other Names: Lexapro; escitalopram; Prozac; fluoxetine; Sertraline; Zoloft
  Arms: SSRIs
Behavioral: CBT — Cognitive Behavior Therapy: 40 patients will receive 16- 20 60 minute sessions of procedurally determined Cognitive Therapy (Beck, 1979) over 14 weeks. Patients will begin with 2 sessions per week which may be reduced to once per week in the latter part of the study period if the patient is responding to the therapy. Cognitive Therapy is designed to teach skills that help to reduce depressive severity. Each session will be videotaped and will include homework to be completed and brought to the following session.
  Other Names: CT; Cognitive Therapy
  Arms: CBT

SUMMARY:
Our goals are 1) to use functional magnetic resonance imaging (fMRI) to predict which depressed individuals will respond to different validated treatments for unipolar depression including Cognitive Therapy (CT) and antidepressant medications (selective serotonin reuptake inhibitors; SSRIs) and 2) to understand whether CT and SSRIs affect similar aspects of brain function underlying cognition and emotion. Thus, we will examine depressed adults ages 18-55 using fMRI during cognitive and emotional information processing tasks, before and after treatment with an SSRI (n=25) or CT (n=40). We hypothesize that: 1) Recovery will occur in treatment with an SSRI primarily for individuals with increased reactivity in limbic brain regions associated with emotion generation and prefrontal regions associated with regulation,. 2) Recovery with CT will occur for patients with increased activity in brain regions associated with emotion generation but decreased activity in prefrontal regions associated with emotion regulation. 3) Recovery with an SSRI will yield similar changes in brain function to CT in brain regions associated with emotion generation but less change in brain regions responsible for emotion regulation such as the prefrontal cortex. Findings from this study may have a profound impact on reducing the burden of clinical depression by providing evidenced-based diagnostic and treatment guidelines.

DETAILED DESCRIPTION:
Same as above.

ELIGIBILITY:
Inclusion Criteria:

1. Meet Diagnostic and Statistical Manual-IV criteria for major depressive disorder (one or more lifetime episodes, separated by at least two months of a return to normal functioning, in a current episode).
2. Male or female outpatients between the ages of 18 and 55 at time of enrollment.
3. Females only must be surgically sterile, post-menopausal for at least one year, or not pregnant and using a method of birth control that is acceptable to the investigator.
4. Have a total score of 14 or more on the first 17-items of the Hamilton Rating Scale for Depression at both the initial and secondary interviews.
5. Be in reasonably good health. Patients with hypothyroidism, diabetes, high blood pressure, chronic respiratory, or other medical conditions may be considered candidates for study enrollment at the discretion of the investigator if their conditions are stable, they have been receiving standard therapies for the treatment of the condition, the prescribed dose and regiment of medication has been stable for at least 3 months, and all appropriate clinical and lab parameters are within normal limits for the condition that are clinically acceptable to the investigator
6. Be free of prescription psychotropic medications for two weeks (four weeks for fluoxetine) before study entry.
7. Provide written informed consent

Exclusion Criteria:

1. Being unable to complete questionnaires written in English, representing an active suicide risk (see below), active alcohol or drug dependence, having any eye problems or difficulties in corrected vision, having a North American Adult Reading Test (NAART) equivalent Full Scale Intelligence Quotient < 85.
2. Pregnant women and those planning to become pregnant during the first 11 months after intake will also be excluded from the study. Pregnancy will be determined by self-report at the interview and by a pregnancy test at the time of the Magnetic Resonance Imaging scan. There will be no cost to the participant for the pregnancy test.
3. People who have metallic foreign objects in their body, such as aneurysm clips or pacemakers, as well as individuals prone to panicking in enclosed spaces will be excluded from the study. Subjects with a questionable history of metallic fragments will also be excluded.
4. Participants who are taking psychotropic medications, particularly antidepressant medications within two weeks of study entry (4 weeks for fluoxetine) will be excluded.
5. Participants will not be excluded on the basis of herbs, supplements, and other prescription or over the counter drugs other than those noted. HIV serostatus will not be evaluated for the research study.
6. At the initial screening visit, if girth seems to present a potential issue for the MRI, than width of participant will be assessed using a hula-hoop that is approximately the same diameter as the MRI scanner. If subject exceeds the width of the hula-hoop, then they will be excluded from the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2008-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Treatment outcome will be assessed on a variety of dimensions including change in symptoms, self-reported rumination, behavioral performance on cognitive tasks, and physiological reactivity to emotional information processing tasks. | 14-16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Greg J Siegle, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Mood Disorders Treatment and Research Program - UPMC, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Siegle GJ, Carter CS, Thase ME. Use of FMRI to predict recovery from unipolar depression with cognitive behavior therapy. Am J Psychiatry. 2006 Apr;163(4):735-8. doi: 10.1176/ajp.2006.163.4.735. PMID 16585452
- [Result] Siegle GJ, Thompson WK, Collier A, Berman SR, Feldmiller J, Thase ME, Friedman ES. Toward clinically useful neuroimaging in depression treatment: prognostic utility of subgenual cingulate activity for determining depression outcome in cognitive therapy across studies, scanners, and patient characteristics. Arch Gen Psychiatry. 2012 Sep;69(9):913-24. doi: 10.1001/archgenpsychiatry.2012.65. PMID 22945620
- [Result] Horner MS, Siegle GJ, Schwartz RM, Price RB, Haggerty AE, Collier A, Friedman ES. C'mon get happy: reduced magnitude and duration of response during a positive-affect induction in depression. Depress Anxiety. 2014 Nov;31(11):952-60. doi: 10.1002/da.22244. Epub 2014 Mar 18. PMID 24643964
- See also: Program in Cognitive Affective Neuroscience website — http://www.wpic.pitt.edu/research/pican/
- See also: PI website — http://www.pitt.edu/~gsiegle/